CLINICAL TRIAL: NCT05856175
Title: The Recurrence Mechanism of Venous Tinnitus After Boney Wall Reconstruction Based on Multimodal Imaging and Multiphysics Coupling
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wang, Zhenchang, Vice President, Director of Medical Imaging Center, Beijing Friendship Hospital
Other Study IDs: 202304
Record Dates: First submitted 2023-04-24; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Pulsatile Tinnitus
Keywords: magnetic resonance angiography; head and neck; ear; pulsatile tinnitus; hemodynamics
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PT patients with postoperative recurrence: participants in this group undergo ultra-high resolution CT, vessel wall MR, 4D Flow MR and ASL MR imaging technology before and after surgery.
- PT patients without postoperative recurrence: participants in this group undergo ultra-high resolution CT, vessel wall MR, 4D Flow MR and ASL MR imaging technology before and after surgery.

SUMMARY:
Venous tinnitus (VT) is seriously affecting the quality of life of five million patients in China. Bony wall reconstruction is the main treatment method, but the postoperative recurrence rate exceeds 30%, and the specific mechanism is unclear. Based on our previous work, a scientific hypothesis was put forward: the key to the recurrence of V T is pathologic remodeling of the peri-sinus bony wall mediated by the venous sinus morphology, blood flow, and pressure after surgical reconstruction. As a continuation of the National Natural Science Foundation of China-Youth Project, this project intends to combine multimodal imaging technology, multiphysics coupled numerical model and machine learning method to analyze analyze the data after bone wall reconstruction in multiple dimensions: ① To explore the influence of peri-sinus bony wall morphology, venous sinus morphology, intra-sinus blood flow, intra-sinus pressure, and cerebral perfusion on the recurrence of VT using ultra-high resolution CT, vessel wall MR, 4D Flow MR and ASL MR imaging technology; ② To explore the influence of blood flow impact, sinus wall pressure and peri-sinus bone wall deformation on the recurrence of VT using multiphysics coupling numerical model with vessel, blood flow, bone and acoustic fields; ③ To determine the risk factors and their weights of VT recurrence using machine learning methods, and to establish a personalized surgical planning and prognostic evaluation models; Thus, to verify the hemodynamic and biomechanical mechanisms of VPT recurrence to achieve personalized and effectively treatment. This project may prevent and warn the recurrence of VPT after bony wall reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* patients with venous tinnitus, a rhythmic noise that follows the heart beating without external stimuli and can disappear or significantly reduce after compression of the affected side of the neck
* the normal otoscopy
* venous tinnitus patients with confirmed sigmoid sinus wall dehiscence with or without sigmoid sinuses enlargement, diverticula and transverse sinuses stenosis using dual-phase enhanced CT examination
* preoperative DSA examination
* bone wall reconstruction

Exclusion Criteria:

* contraindications for CT and MR Examination
* tumor and arterial abnormalities

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * postoperative recurrence patients：100 cases
  * no postoperative recurrence patients：50 cases
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
the influence of peri-sinus bony wall morphology on the recurrence of pulsatile tinnitus using CT | 2023.6.1-2025.12.31
  ultra-high resolution CT
the influence of venous sinus morphology, intra-sinus blood flow, and intra-sinus pressure on the recurrence of pulsatile tinnitus using MRI | 2023.6.1-2025.12.31
  4D Flow MR imaging technology
the influence of cerebral perfusion on the recurrence of pulsatile tinnitus using MRI | 2023.6.1-2025.12.31
  ASL MR imaging technology
the influence of blood flow impact, sinus wall pressure and peri-sinus bone wall deformation on the recurrence of pulsatile tinnitus | 2023.6.1-2025.12.31
  multiphysics coupling numerical model with vessel, blood flow, bone and acoustic fields
the risk factors and their weights of pulsatile tinnitus recurrence | 2023.6.1-2025.12.31
  Ensight, a post-processing software, was used to study the interaction between hemodynamic features and acoustic features with multivariate analysis and machine learning methods.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenchang Wang, Prof., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
the project team has not decided the ways to share the data